CLINICAL TRIAL: NCT04948320
Title: Temporomandibular Dysfunction Affects Neck Disability, Headache, Anxiety, And Sleep Quality In Women: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, sevilay seda bas, Research assistant, Ankara Yildirim Beyazıt University
Other Study IDs: 2020-43
Record Dates: First submitted 2021-06-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Temporomandibular Disorders; Headache; Neck Disorder; Anxiety; Sleep Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders; Headache; Anxiety Disorders; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temporomandibular Disorder Group
- Control Group

SUMMARY:
The temporomandibular joint (TMJ), is the only movable joint between the joints in the head and neck system. It is a component of the chewing system and is involved in important functions such as speech, swallowing, taste and breathing. Temporomandibular dysfunction (TMD) is the general name given to various musculoskeletal problems seen in the stomatognathic system, mostly affecting the masticatory muscles and/or TMJ. TMD is the second most common musculoskeletal pain after chronic low back pain. Patients with TMD may also complain of other musculoskeletal problems, craniocervical problems, sleep problems, and anxiety disorders. The aim of this study is to investigate, compare and examine the relationship between neck dysfunction, headache and temporomandibular dysfunction severity, anxiety and sleep quality in female individuals.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years
* Temporomandibular disorders more than 6 months
* Volunteering

Exclusion Criteria:

* Cranio-cervical trauma and temporomandibular operation history
* Infection
* 20-40 points from Fonseca Anamnestic Index 20-40 points

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: temporomandibular disorder and healthy women
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline

SECONDARY OUTCOMES:
Fonseca Anamnestic Index | Baseline
Numerical Rating Scale | Baseline
Neck Disability Index | Baseline
Headache Impact Test | baseline
General Anxiety Disorder-7 Scale | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No